CLINICAL TRIAL: NCT03121547
Title: Opioid Induced Gait Variability
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Henning Bliddal, Professor, Frederiksberg University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 131
Record Dates: First submitted 2017-04-10; First posted 2017-04-20 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Opioid Induced Motor Disturbances
MeSH Terms: interventions — Tapentadol; Tablets; Tramadol; Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo oral tablet (Placebo Comparator): One inert calcium tablet is administered after a set of baseline measurements are performed. Subsequently outcomes are assessed every hour for 6 hours, yielding a total of 7 hourly measurements.
  Interventions: Drug: Placebo Oral Tablet
- Tramadol Hydrochloride 100 mg Extended Release Oral Tablet (Experimental): One tablet containing 100 milligrams (mg) Mandolgin Retard, Sandoz is administered after a set of baseline measurements are performed. Subsequently outcomes are assessed every hour for 6 hours, yielding a total of 7 hourly measurements.
  Interventions: Drug: Tramadol Hydrochloride 100 mg Extended Release Oral Tablet
- Tapentadol 50 mg Oral Tablet (Experimental): One tablet containing 50 milligrams (mg) Palexia Depot, Grünenthal is administered after a set of baseline measurements are performed. Subsequently outcomes are assessed every hour for 6 hours, yielding a total of 7 hourly measurements.
  Interventions: Drug: Tapentadol 50 mg Oral Tablet

INTERVENTIONS:
Drug: Tapentadol 50 mg Oral Tablet — 1 tablet administered
  Other Names: Palexia Depot (50 mg)
  Arms: Tapentadol 50 mg Oral Tablet
Drug: Tramadol Hydrochloride 100 mg Extended Release Oral Tablet — 1 tablet administered
  Other Names: Mandolgin Retard (100 mg)
  Arms: Tramadol Hydrochloride 100 mg Extended Release Oral Tablet
Drug: Placebo Oral Tablet — calcium tablet
  Other Names: Calcium tablet
  Arms: Placebo oral tablet

SUMMARY:
While the analgesic effects of opioids are well known, evidence suggest that there are differences in the adverse dizziness of the different opioid types, which may influence the gait function differently. However, this has not been investigated scientifically under controlled conditions. Normal gait function is characterized by cyclic movements with a high degree of predictability. As such, the amount of kinematic variability can provide important information about a condition or an intervention that may affect the gait function . Three-dimensional gait analysis is a recognized method to assess changes in stride-to-stride variability associated with a medical condition or caused by an intervention. Thus, opioid induced changes in gait variability, and possible differences between opioid types, can be assessed objectively from differences in the variability of movements obtained from a three-dimensional gait analysis.

The purpose of this study is to investigate differences in gait variability induced by two different single-dose opioid formulations and an inert placebo in healthy volunteers and knee osteoarthritis patients.

DETAILED DESCRIPTION:
The study is designed as an experimental single center, double-blind treatment, cross-over study with inert placebo, Tapentadol (Palexia Depot), and Tramadolhydrochlorid (Mandolgin Retard), with a minimum of 7days wash-out periods.

At day 1 (Visit 1), baseline measurements are carried out before tablet administration. Immediately after baseline measurements one tablet is administered, and hourly measurements are performed for 6 hours. Subsequently all participants enter a minimum 7 day washout period, after which they return to the facility to repeat the procedures at Visit 2 (day 8+) and Visit 3 (day 15+). The order of treatments will be randomized (1:1:1).

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects:

* In general good health, in the opinion of the Investigator, based on medical history and physical examination.
* Ability to comprehend and a willingness to provide written informed consent
* Age between 50 and 75 years
* No opioid usage 3 months prior to the study
* No musculoskeletal pain requiring medical attention during the previous 3 months
* Willing and able to complete study visits and procedures
* Willing to hold activity, exercise level, and concurrent treatments/therapies generally consistent during the study
* A body mass index (BMI) of ≤30

Patients with knee osteoarthritis (OA)

* Diagnosis of knee OA
* Ability to comprehend and a willingness to provide written informed consent
* Age between 50 and 75 years
* No opioid usage 3 months prior to the study
* Knee pain of at least 40 mm on a 0-100 mm visual analog scale (without analgesics) representing the average pain intensity during the previous week
* Willing to discontinue all pain medications 24 hours before and during examination visits
* Willing and able to complete study visits and procedures
* Willing to hold activity, exercise level, and concurrent treatments/therapies generally consistent during the study
* In general good health, in the opinion of the Investigator, based on medical history and physical examination.
* A body mass index (BMI) of ≤30

Exclusion Criteria:

The same exclusion criteria apply for both healthy subjects and patients with knee osteoarthritis:

* Clinical signs of gait ataxia assessed by clinical neurological examination
* Independent or unsteady walking (i.e. dependence on walking device or stumbling gait)
* Counter indications to either of the investigational products, including but not restricted to:

  * Allergy towards one or more of the investigational products or their excipient(s).
  * Significant respiratory depression
  * Current or serious asthma
  * Hypercapnia
  * Suspected or diagnosed paralytic ileus
  * Acute intoxication by alcohol, hypnotica, centrally acting analgesics, psychopharmaca or other pharmaceuticals.
  * Renal dysfunction
  * Hepatic dysfunction
  * Diseases of the biliary tract
  * Acute pancreatitis
  * Usage of monoamine oxidase inhibitors within the last 14 days
  * Galactose intolerance
  * Lactase deficiency
  * Glucose/galactose malabsorption
  * Epilepsy
* Previous usage of opioids without pain reliving effect.
* Patients who have a documented history of an allergic reaction or a clinically significant intolerance to opioids
* Malignant pain
* Excessive joint laxity in the lower extremities indicative of functional ligamentous deficiency.
* Dependency of walking aid (stick, cane, roller etc.).
* Positive Clock Drawing Test
* Abuse of alcohol, medicine and narcotics within past 5 years.
* History of symptoms of autoimmune disorders
* Diabetes
* Pregnancy or breast feeding
* History, diagnosis, or signs and symptoms of clinically significant neurological disease
* History, diagnosis, signs or symptoms of any clinically significant psychiatric disorder

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05-19 (Actual); Primary Completion 2016-01-29 (Actual); Study Completion 2016-01-29 (Actual)

PRIMARY OUTCOMES:
Changes in Gait variability | every hour from pre-tablet administration (hour 0) to hour 6
  Three dimensional gait analysis during 6 minutes of continuous treadmill walking.

SECONDARY OUTCOMES:
Self reported dizziness | every hour from pre-tablet administration (hour 0) to hour 6
  Current dizziness is assessed by means of a 100 mm visual analog scale
Self reported knee pain | every hour from pre-tablet administration (hour 0) to hour 6
  Current knee pain is assessed by means of a 100 mm visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bliddal, DMSc, Principal Investigator — The Parker Institute
Locations (1):
- The Parker Institute, Frederiksberg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Henriksen M, Alkjaer T, Raffalt PC, Jorgensen L, Bartholdy C, Hansen SH, Bliddal H. Opioid-Induced Reductions in Gait Variability in Healthy Volunteers and Individuals with Knee Osteoarthritis. Pain Med. 2019 Nov 1;20(11):2106-2114. doi: 10.1093/pm/pny286. PMID 30649458